CLINICAL TRIAL: NCT04872322
Title: Randomized Study of the Effect of Initial Ropivacaine Dosage During Continuous Popliteal Nerve Blocks on Rebound Pain in Foot and Ankle Surgery
Brief Title: Effect of Ropivacaine During Popliteal Nerve Block in Foot and Ankle Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRAI17D.481
Record Dates: First submitted 2021-05-03; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Popliteal Nerve Block; Foot Surgery; Ankle Surgery
MeSH Terms: interventions — Ropivacaine; oxycodone-acetaminophen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Popliteal Nerve Block (Active Comparator): Participants undergoing foot or ankle surgery will receive an initial injection of 0.5% ropivacaine as the initial anesthetic followed by continuous injection of 0.25% ropivacaine.
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution; Drug: Ropivacaine 0.25% Injectable Solution; Drug: Percocet Pill; Drug: Norco Pill; Procedure: Foot/Ankle Surgery
- Partial Popliteal Nerve Block (Active Comparator): Participants undergoing foot or ankle surgery will receive 0.25% ropivacaine initially followed by the usual continuous injection of 0.25% ropivacaine during surgery
  Interventions: Drug: Ropivacaine 0.25% Injectable Solution; Drug: Percocet Pill; Drug: Norco Pill; Procedure: Foot/Ankle Surgery

INTERVENTIONS:
Drug: Ropivacaine 0.5% Injectable Solution — Participants will receive the nerve block preoperatively using 0.5% ropivacaine
  Arms: Standard Popliteal Nerve Block
Drug: Ropivacaine 0.25% Injectable Solution — Participants will receive the nerve block preoperatively using 0.25% ropivacaine
Drug: Percocet Pill — After surgery participants will be given a prescription for Percocet to be taken as needed for pain
Drug: Norco Pill — After surgery participants will be given a prescription for Norco to be taken as needed for pain
Procedure: Foot/Ankle Surgery — Participant will undergo foot or ankle surgery and receive a popliteal nerve block

SUMMARY:
With the increasing rise of outpatient surgery in orthopaedic procedures, the management of immediate postoperative pain has been a major topic investigated, with the use of a peripheral nerve block in combination with general anesthesia being a commonly accepted method. Foot and ankle procedures, which offer the choice of several anesthetic techniques, have increasingly been performed with this method predominantly through the combination of general anesthesia with a single-injection popliteal nerve block to reduce the substantial acute postoperative pain that often requires large opioid intake within the post-anesthesia care unit (PACU). However, as a single-injection peripheral nerve block resolves off shortly following surgery, major postoperative pain, termed "rebound pain", can also arise, and has the potential to be even greater than that of patients who do not receive any peripheral nerve block with general anesthesia.

The purpose of this study is to evaluate the contribution of ropivacaine concentration (0.5% versus 0.25%) of the initial bolus in continuous popliteal nerve blocks toward the rebound pain phenomena, or the quantifiable difference in pain experienced during the initial time after block resolution, in foot and ankle surgeries.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing foot and ankle surgeries under the care of Dr. Steven Raikin with continuous popliteal blocks at Riverview Surgical Center will be considered for enrollment.

Exclusion Criteria:

* Patients who present with a) known hypersensitivity to ropivacaine or to any local anesthetic agent of the amide type,
* Existing use of narcotics,
* Pregnant women,
* Individuals under the age of 18
* Procedures involving any other forms of anesthesia other than general anesthesia with a continuous popliteal nerve block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2017-08-31 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | 7 days
  Participants Satisfaction with pain control will be measured using the Visual Analog Scale for Pain (VAS)
Postoperative Opioid Usage | 7 days
  For each group, participants will be asked to record their postoperative pain medication usage daily

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States